CLINICAL TRIAL: NCT05262985
Title: Durvalumab (MEDI4736) Plus Platinum-based Chemotherapy in Advanced LCNEC: a Pilot Phase II Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Elizabeth Dudnik (Other)
Responsible Party: Sponsor-Investigator, Elizabeth Dudnik, Dr. Elizabeta Dudnik, Assuta Medical Center
Organization: Assuta Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-20-20907
Record Dates: First submitted 2022-02-20; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Patients With Advanced Treatment Naive LCNEC
MeSH Terms: interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with Durvalumab+ (Other): Comparison of standard treatment verses the addition of Durvalomab to the standard protocol.
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — In patients with advanced treatment naive LCNEC, treatment with Durvalumab+ Cisplatin/Carboplatin+Etoposide

SUMMARY:
PROTOCOL SYNOPSIS Clinical Protocol ESR-20-20907 Study Title: Durvalumab (MEDI4736) plus platinum-based chemotherapy in advanced large-cell neuroendocrine tumors of lung (LCNEC): a pilot phase II study Protocol Number: ESR-20-20907 Clinical Phase: phase II Study Duration: 30 months

Investigational Product(s) and Reference Therapy:

Investigational Product: Durvalumab (MEDI4736) Durvalumab concentrate for solution for infusion will be supplied in glass vials containing 500 mg durvalumab at a concentration of 50 mg/mL Reference Therapy: Cisplatin/Carboplatin+Etoposide Research Hypothesis

Primary hypothesis:

1.1 In patients with advanced treatment naive LCNEC, treatment with Durvalumab+ Cisplatin/Carboplatin+Etoposide is associated with 12-month PFS rate of at least 18%.

Secondary hypothesis:

1.2 In patients with advanced treatment naïve LCNEC, treatment with Durvalumab+ Cisplatin/Carboplatin+Etoposide is associated with ORR of 50%.

1.3 In patients with advanced treatment naïve LCNEC, treatment with Durvalumab+ Cisplatin/Carboplatin+Etoposide is associated with 12-months OS rate of at least 50%.

1.4 Incidence of grade ≥3 adverse events is less than 60%.

Exploratory hypothesis:

1.5 There is a positive correlation between the small-cell lung cancer-like molecular subtype and efficacy parameters (ORR, PFS, OS), and also between high TMB and efficacy parameters (ORR, PFS, OS) of treatment with Durvalumab+Cisplatin/Carboplatin+Etoposide in patients with advanced treatment naive LCNEC.

Objectives

Primary Objective:

1.1 To assess progression-free survival (PFS at 12 months, RECIST v. 1.1) with Durvalumab+ Cisplatin/Carboplatin+Etoposide in patients with advanced treatment-naive LCNEC.

Secondary Objectives:

1.2 To assess objective response rate (ORR at best response) according to Response Evaluation Criteria in Solid Tumors, v. 1.1 (RECIST v. 1.1) with Durvalumab+ Cisplatin/Carboplatin+Etoposide in patients with advanced treatment naive LCNEC.

1.3 To assess overall survival (OS at 12 months) with Durvalumab+ Cisplatin/Carboplatin+Etoposide in patients with advanced treatment-naive LCNEC.

1.4 To further evaluate the safety profile of Durvalumab+Cisplatin/Carboplatin+Etoposide in patients with advanced treatment naive LCNEC (CTCAE v. 5.0).

Exploratory Objectives:

1.5 To assess the predictive effect of tumor molecular subtype (small-cell lung cancer - like versus non-small cell lung cancer - like, assessed by NGS), tumor mutational burden (TMB, mut/Mb assessed by NGS) and PD-L1 (assessed by TPS - by IHC using 22C3 antibody) on ORR, PFS, and OS with Durvalumab+Cisplatin/Carboplatin+Etoposide in patients with advanced treatment-naive LCNEC.

Study Design:

* Open-label non-randomized non-comparative single-center pilot phase 2 study
* Response assessment: brain/chest/abdominal/pelvic CT scan every 8 weeks+-7 days
* PFS, ORR - assessed by the board-certified radiology expert experienced in RECIST v. 1.1 evaluation; OS assessment

Number of Centers: single center Number of Patients: 22

Study Population:

Adult patients (aged ≥18 years) with histologically or cytologically documented advanced LCNEC (stage IV or stage III not eligible for definitive treatment) without prior systemic treatment for advanced disease.

Investigational Product(s), Dose and Mode of Administration:

The enrolled patients will receive IV durvalumab 1500 mg (administered on day 1 of each 21-day cycle), IV etoposide 100 mg/m² (administered on days 1-3 of each 21-day cycle), with investigator's choice of either IV carboplatin area under the curve 5 mg/mL per min or IV cisplatin 80 mg/m² (administered on day 1 of each 21-day cycle) for four cycles followed by maintenance IV durvalumab 1500 mg (administered on day 1 of each 28-day cycle).

ELIGIBILITY:
Inclusion Criteria:

* Advanced- stage (stage IV or stage III not eligible for definitive treatment) LCNEC without prior systemic treatment for advanced disease

  * Measurable disease by RECIST 1.1 criteria (at least 1 lesion, not previously irradiated, that qualifies as a RECIST 1.1 target lesion (TL) at baseline)
  * ECOG PS≤1
  * Body weight >30kg
  * Life expectancy of at least 3 months
  * Brain metastases are allowed providing these are asymptomatic or clinically stable after surgery or radiation therapy (either stereotactic radiotherapy or whole brain radiotherapy), and not requiring corticosteroid therapy

    - 10 mg prednisone or equivalent are allowed
  * Normal hematologic, renal, liver and thyroid function parameters:

    * Absolute neutrophil count ≥ 1500/mm3, platelets ≥ 100,000/mm3, hemoglobin ≥ 9 g/dL;
    * Creatinine clearance ≥ 40 mL/min (≥ 50 mL/min if cisplatin-based regimen will be chosen);
    * Total bilirubin ≤ 1.5 mg/dL; ALT+ AST levels £ 2.5 × ULN; for patients with liver metastases £ 5 × ULN;
  * TSH within normal limits, if TSH is abnormal - normal total T3/free T3 and free T4
  * Female patients with reproductive potential (postmenopausal: ≥ 12 months of non-therapy-induced amenorrhea or surgically sterile) must have a negative pregnancy test (serum/urine) prior to starting treatment
  * All female patients with reproductive potential and male patients with partners of childbearing potential, must agree to use barrier contraception methods while receiving the study treatment and for 90 days after stopping the study treatment
  * Age ≥18
  * Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations
  * Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow-up

Exclusion Criteria:

* Exclusion Criteria:

  * Carcinomatous meningitis or history of carcinomatous meningitis
  * Prior treatment with an anti-PD-1/anti-PD-L1 agent/chemotherapy
* Patients who have received prior anti-PD-1/anti-PD-L1 agent/platinum-based chemotherapy as neo-adjuvant or adjuvant therapy with curative intent for non-metastatic disease must have experienced a disease-free interval of at least 6 months since the last anti-PD-1/anti-PD-L1 agent/chemotherapy administration.

  • Patients who have received prior anti-PD-1/anti-PD-L1 agent:
* Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
* All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study
* Must not have experienced a ≥Grade 3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy; patients with endocrine AE of ≤Grade 2 are permitted to enrol if they are stably maintained on appropriate replacement therapy and are asymptomatic
* Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day

  • Any unresolved toxicity ≥Grade 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria:
* Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consulting PI
* Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consulting PI

  • Radiation therapy to the brain/lung within 1 week of study treatment
* Prior radiation to other sites (excluding brain and lung) may be completed at any point prior to study treatment

  * Major surgery within 4 weeks of study treatment
  * Any concurrent chemotherapy (other than per protocol), immune check-point inhibitors, biologic, or hormonal therapy for cancer treatment
  * Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:
* Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
* Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
* Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)

Receipt of live attenuated vaccine within 30 days prior to the study treatment initiation; if enrolled, patients should not receive live vaccine whilst receiving study treatment and up to 30 days after the last dose of study treatment

* Body weight<30 kg
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], systemic lupus erythematosus, sarcoidosis, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included on an individual basis after consulting PI
  * Patients with celiac disease controlled by diet alone
* Prior allogeneic bone marrow transplantation or solid organ transplant
* History of active primary immunodeficiency
* AIDS/HIV positivity (by history)
* Active tuberculosis
* Patients with active hepatitis B (HBV, chronic or acute; defined as having a positive hepatitis B surface antigen (HBsAg) test at screening) or hepatitis C

  * Patients with past HBV infection or resolved HBV infection (defined as the presence of hepatitis B core (HBc) antibody and absence of HBsAg) are eligible
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA
* Any evidence of severe or uncontrolled concurrent condition that places patient at an unacceptable risk from participation in the study/confounds the ability to interpret study data, limits compliance with study requirements, substantially increases the risk of incurring AEs, including but not limited to active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, chronic diarrhea, interstitial lung disease
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of study treatment and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* Contraindication for CT
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy
* Inability to sign the informed consent form
* Concurrent enrolment in another clinical study unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study more than 4 weeks since last study treatment
* Prior randomization or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
To assess progression-free survival (PFS at 12 months, RECIST v. 1.1) with Durvalumab+ Cisplatin/Carboplatin+Etoposide in patients with advanced treatment-naive LCNEC | At 12 months

SECONDARY OUTCOMES:
To assess objective response rate (ORR at best response) according to Response Evaluation Criteria in Solid Tumors, v. 1.1 (RECIST v. 1.1) with Durvalumab+ Cisplatin/Carboplatin+Etoposide in patients with advanced treatment naive LCNEC. | At 12 months
To assess overall survival (OS at 12 months) with Durvalumab+ Cisplatin/Carboplatin+Etoposide in patients with advanced treatment-naive LCNEC. | At 12 months
To further evaluate the safety profile of Durvalumab+Cisplatin/Carboplatin+Etoposide in patients with advanced treatment naive LCNEC (CTCAE v. 5.0). | At 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assuta MC, Tel Aviv, Israel